CLINICAL TRIAL: NCT02038842
Title: Phase I/II Open-label Randomized Multicenter Trial to Assess Immunogenicity and Safety of 4 Prime-boost Combinations of HIV Vaccine Candidates (MVA HIV-B/LIPO-5; LIPO-5/MVA HIV-B; GTU®-MultiHIV B/LIPO-5; GTU®-MultiHIV B/MVA HIV-B) in Healthy Volunteers at Low Risk of HIV Infection
Brief Title: Immunogenicity and Safety of 4 Prime-boost Combinations of HIV Vaccine Candidates in Healthy Volunteers
Acronym: VRI01
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012-002456-17
Record Dates: First submitted 2014-01-02; First posted 2014-01-17 (Estimated); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MVA HIV-B and LIPO-5 vaccines (Experimental): MVA HIV-B primes 0,5 milliliter (mL) Intramuscular at Week 0 and Week 8 LIPO-5 1mL Intramuscular boosts at Week 20 and Week 28
  Interventions: Biological: LIPO-5; Biological: MVA HIV-B (MVATG17401)
- LIPO-5 and MVA HIV-B vaccines (Experimental): LIPO-5 primes 1mL intramuscular at Week 0 and Week 8 and MVA HIV-B 0,5mL intramuscular boosts at Week 20 and Week 28
  Interventions: Biological: LIPO-5; Biological: MVA HIV-B (MVATG17401)
- GTU-MultiHIV B and LIPO-5 vaccines (Experimental): GTU-MultiHIV B 0,5mL intramuscular via Biojector 2000 and 0,5mL intradermic primes at Week 0, Week 4 and Week 12 and LIPO-5 1mL intramuscular boosts at Week 20 and Week 28
  Interventions: Biological: LIPO-5; Biological: GTU®-MultiHIV B: 0.5 mL IM via Biojector® 2000 and 0.5mL IntraDermic, 3 shots
- GTU-MultiHIV B and MVA HIV-B vaccines (Experimental): GTU-MultiHIV B 0,5mL intramuscular via Biojector 2000 and 0,5mL intradermic primes at Week 0, Week 4 and Week 12 and MVA HIV-B 0,5mL intramuscular boosts at Week 20 and Week 28
  Interventions: Biological: MVA HIV-B (MVATG17401); Biological: GTU®-MultiHIV B: 0.5 mL IM via Biojector® 2000 and 0.5mL IntraDermic, 3 shots

INTERVENTIONS:
Biological: LIPO-5 — LIPO-5: 1mL IntraMuscular, 2 shots;
  Other Names: ANRS LIPO-5 vaccine candidate; ANRS MVA HIV-B (MVATG17401) vaccine candidate; FIT Biotech GTU-MultiHIV B vaccine candidate
  Arms: GTU-MultiHIV B and LIPO-5 vaccines; LIPO-5 and MVA HIV-B vaccines; MVA HIV-B and LIPO-5 vaccines
Biological: MVA HIV-B (MVATG17401) — MVA HIV-B (MVATG17401): 0.5mL IntraMuscular, 2 shots;
  Arms: GTU-MultiHIV B and MVA HIV-B vaccines; LIPO-5 and MVA HIV-B vaccines; MVA HIV-B and LIPO-5 vaccines
Biological: GTU®-MultiHIV B: 0.5 mL IM via Biojector® 2000 and 0.5mL IntraDermic, 3 shots — GTU®-MultiHIV B: 0.5 mL IM via Biojector® 2000 and 0.5mL IntraDermic, 3 shots
  Arms: GTU-MultiHIV B and LIPO-5 vaccines; GTU-MultiHIV B and MVA HIV-B vaccines

SUMMARY:
The development of a safe and effective HIV-1 vaccine strategy would probably be the best solution for the ultimate control of the worldwide AIDS pandemic. Heterologous prime-boost immunisations are today considered promising HIV prophylactic vaccine strategies. It is thus relevant to pursue the development of different candidate vaccines in prime-boost vaccine strategies to identify the most promising prime-boost combinations and to integrate scientific inquiry into trial protocols from the beginning to maximize learning opportunities.

DETAILED DESCRIPTION:
Phase I/II, multicenter, national, open-label, randomized trial HIV including 4 prophylactic prime-boost HIV vaccines strategies:

Volunteers are randomly allocated in a 1:1:1:1 ratio at trial entry to 4 parallel arms with the following prime-boost strategies:

Arm 1. MVA HIV-B primes at Week 0 and Week 8 + LIPO-5 boosts at Week 20 and Week 28 Arm 2. LIPO-5 primes at Week 0 and Week 8 + MVA HIV-B boosts at Week 20 and Week 28 Arm 3. GTU-MultiHIV B primes at Week 0, Week 4 and Week 12 + LIPO-5 boosts at Week 20 and Week 28 Arm 4. GTU-MultiHIV B primes at Week 0, Week 4 and Week 12 + MVA HIV-B boosts at Week 20 and Week 28

ELIGIBILITY:
Inclusion Criteria:

* Written and signed informed consent
* Subject at low risk to contract HIV i.e.

  * no history of injecting drug use in the previous ten years;
  * no gonorrhea or syphilis in the last six months;
  * no high risk partner (e.g. injecting drug user, HIV positive partner) either currently or within the past six months ;
  * no unprotected anal intercourse in the last six months, outside a relationship with a regular partner known/presumed to be HIV negative ;
  * no unprotected vaginal intercourse in the last six months outside a relationship with a regular known/presumed HIV negative partner
* Available for follow-up for the duration of the study (56 weeks from screening)
* Willing to undergo a HIV test
* Willing to undergo a genital infection screen
* If heterosexually active female, using an effective method of contraception with partner (combined oral contraceptive pill; injectable contraceptive; contraceptive implant/patch; IntraUterine Contraceptive Device (IUCD); consistent record with condoms if using these; physiological or anatomical sterility in self or partner) from 14 days prior to the first vaccination until 4 months after the last, and willing to undergo urine pregnancy tests prior to each vaccination
* If heterosexually active male, using an effective method of contraception with their partner from the first day of vaccination until 4 months after the last vaccination
* Subject registered in French Health ministry computerised file and authorised to participate in a clinical trial
* Subject covered by Health Insurance

Exclusion Criteria:

* Clinically relevant abnormality on history or examination including history of:

  * uncontrolled infection;
  * autoimmune disease;
  * immunodeficiency or use of immunosuppressive drugs within 3 months prior to screening;
  * cancer;
  * chronic diseases requiring long-term treatment whose interruption during the trial has no impact on the health status in the short or long-term
* Receipt of live attenuated vaccine within 60 days or other vaccine within 14 days prior to W0
* Planned receipt of other vaccines than those planned by the protocol and those recommended in France (excluding live attenuated vaccines) during the trial follow-up (reference : Weekly Epidemiological Newsletter 14-15 dated on April 10th, 2012 (Bulletin Epidémiologique hebdomadaire 14-15 / 10 avril 2012))
* Receipt of blood products or immunoglobin within 4 months prior to screening
* History of severe local or general reaction to vaccination defined as

  * local: extensive, indurated redness and swelling involving most of the antero-lateral thigh or the major circumference of the arm, not resolving within 72 hours
  * general: fever ≥ 39.5°C within 48 hours; anaphylaxis; bronchospasm; laryngeal oedema; collapse; convulsions or encephalopathy within 72 hours
* Positive for ANA antibodies at a titer considered clinically significant: titer ≥ local cut-off associated with positive anti-native DNA and extractable nuclear antigen antibodies
* HIV-1 or HIV-2 positive or indeterminate at screening
* Woman expecting to conceive during the study period
* Pregnant or breastfeeding woman
* Symptoms, physical signs or laboratory values suggestive of systemic disorders, including renal, hepatic, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric, which could interfere with the interpretation of the trial results or compromise the health of the volunteers
* Clinically significant grade 1 routine laboratory parameters
* Grade 2 or above routine laboratory parameters
* Known hypersensitivity to aminoglycosides and eggs (as used in the vaccine production processes)
* Known hypersensitivity to one of the trial vaccine components, the metabolites or formulation excipients
* Anticipated non-compliance with the protocol
* Participation in another clinical trial with an on-going exclusion period at screening
* Participation in a HIV preventive vaccine clinical trial (unless participant were randomized in placebo arm)
* Subject under legal guardianship or incapacitation
* Subject who is an active blood donor and unwilling to interrupt blood donations during the his/her participation in the trial

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2014-03; Primary Completion 2015-10 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Daniel LELIEVRE Study Chair, Pr, Principal Investigator — Hopital Henri Mondor; Laura RICHERT Methodologist, Dr, Principal Investigator — Inserm Unit 897
Locations (1):
- Service d'Immunologie Clinique 51, avenue du Marechal de Lattre de Tassigny, Créteil, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteers will be recruited through the ARNS network of volunteers, through advertising via media and through a dedicated website, and given a telephone number to contact.
  From March 2014 to March 2015, 129 participants were screened in four sites in France.
Groups:
- MVA HIV-B/LIPO-5: MVA HIV-B primes 0,5 milliliter (mL) Intramuscular at Week 0 and Week 8 LIPO-5 1mL Intramuscular boosts at Week 20 and Week 28
  LIPO-5: LIPO-5: 1mL IntraMuscular, 2 shots;
  MVA HIV-B (MVATG17401): MVA HIV-B (MVATG17401): 0.5mL IntraMuscular, 2 shots;
- LIPO-5/MVA HIV-B: LIPO-5 primes 1mL intramuscular at Week 0 and Week 8 and MVA HIV-B 0,5mL intramuscular boosts at Week 20 and Week 28
  LIPO-5: LIPO-5: 1mL IntraMuscular, 2 shots;
  MVA HIV-B (MVATG17401): MVA HIV-B (MVATG17401): 0.5mL IntraMuscular, 2 shots;
- GTU-MultiHIV B/LIPO-5: GTU-MultiHIV B 0,5mL intramuscular via Biojector 2000 and 0,5mL intradermic primes at Week 0, Week 4 and Week 12 and LIPO-5 1mL intramuscular boosts at Week 20 and Week 28
  LIPO-5: LIPO-5: 1mL IntraMuscular, 2 shots;
  GTU®-MultiHIV B: 0.5 mL IM via Biojector® 2000 and 0.5mL IntraDermic, 3 shots: GTU®-MultiHIV B: 0.5 mL IM via Biojector® 2000 and 0.5mL IntraDermic, 3 shots
- GTU-MultiHIV B/MVA HIV-B: GTU-MultiHIV B 0,5mL intramuscular via Biojector 2000 and 0,5mL intradermic primes at Week 0, Week 4 and Week 12 and MVA HIV-B 0,5mL intramuscular boosts at Week 20 and Week 28
  MVA HIV-B (MVATG17401): MVA HIV-B (MVATG17401): 0.5mL IntraMuscular, 2 shots;
  GTU®-MultiHIV B: 0.5 mL IM via Biojector® 2000 and 0.5mL IntraDermic, 3 shots: GTU®-MultiHIV B: 0.5 mL IM via Biojector® 2000 and 0.5mL IntraDermic, 3 shots
Period: Overall Study
Arm/Group | MVA HIV-B/LIPO-5 | LIPO-5/MVA HIV-B | GTU-MultiHIV B/LIPO-5 | GTU-MultiHIV B/MVA HIV-B
Started | 23 | 23 | 23 | 23
Completed | 21 | 21 | 18 | 19
Not Completed | 2 | 2 | 5 | 4
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 0
Not completed — Participant decision | 0 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 3 | 1
Not completed — Other (professional impossibility, etc.) | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- MVA HIV-B/LIPO-5: MVA HIV-B primes 0,5mL IntraMuscular at W0 and W8 LIPO-5 1mL IntraMuscular boosts at W20 and W28
- LIPO-5/MVA HIV-B: LIPO-5 primes 1mL IntraMuscular at W0 and W8 MVA HIV-B 0,5mL IntraMuscular boosts at W20 and W28
- GTU-MultiHIV B/LIPO-5: GTU-MultiHIV B 0,5mL IntraMuscular via Biojector 2000 and 0,5mL IntraDermic primes at W0, W4 and W12 LIPO-5 1mL IntraMuscular boosts at W20 and W28
- GTU-MultiHIV B/MVA HIV-B: GTU-MultiHIV B 0,5mL IntraMuscular via Biojector 2000 and 0,5mL IntraDermic primes at W0, W4 and W12 MVA HIV-B 0,5mL IntraMuscular boosts at W20 and W28
- Total: Total of all reporting groups
Arm/Group | MVA HIV-B/LIPO-5 | LIPO-5/MVA HIV-B | GTU-MultiHIV B/LIPO-5 | GTU-MultiHIV B/MVA HIV-B | Total
Number analyzed (Participants) | 23 | 23 | 23 | 23 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 23 | 23 | 23 | 92
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26 [24 to 36] | 24 [22 to 33] | 29 [25 to 38] | 26 [24 to 36] | 27 [24 to 33.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 9 | 14 | 42
  Male | 15 | 12 | 14 | 9 | 50
Region of Enrollment [Number; unit: participants]
  France | 23 | 23 | 23 | 23 | 92

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of the Safety of MVA HIV-B at Week 2 in Arm 1
Description: Count of participants without any grade 3 or 4 adverse events (clinical or biological) related to MVA-vaccine immunisation, reported from Week 0 to Week 2 in arm 1
Time Frame: Visit Week 2
Measure: Count of Participants; unit: Participants
Groups:
- MVA HIV-B/LIPO-5: MVA HIV-B primes 0,5 mL IntraMuscular at W0 and W8 LIPO-5 1mL IntraMuscular boosts at W20 and W28
Arm/Group | MVA HIV-B/LIPO-5
Number analyzed (Participants) | 23
Participants | 22

2. Primary Outcome: To Discard Vaccine Strategies With an Insufficient Level of Immunogenicity, Defined by HIV-specific IFN-γ-ELISPOT Responses, Among 4 HIV Prophylactic Prime-boost Combinations in Healthy Volunteers at Low Risk of HIV Infection
Description: Count of participants with a HIV-specific Interferon-gamma Enzyme Linked Immunosorbent SPOT (IFN-γ ELISPOT) response in each of the 4 arms, defined by a positive response to at least one of the stimulating HIV peptide pools (15-mer pools covering Env, Gag, Pol, and Nef) measured in stimulated Peripheral Blood Mononuclear Cell (PBMC) by a standard IFN-γ ELISPOT assay at Week 30, i.e. 2 weeks after the last vaccine immunisation.
Time Frame: Visit Week 30
Measure: Count of Participants; unit: Participants
Arm/Group | MVA HIV-B/LIPO-5 | LIPO-5/MVA HIV-B | GTU-MultiHIV B/LIPO-5 | GTU-MultiHIV B/MVA HIV-B
Number analyzed (Participants) | 21 | 21 | 19 | 21
Participants | 7 | 9 | 0 | 14
Statistical Analysis 1: Comparison: MVA HIV-B/LIPO-5 vs LIPO-5/MVA HIV-B vs GTU-MultiHIV B/LIPO-5 vs GTU-MultiHIV B/MVA HIV-B; Trial was designed to compare the observed proportion of responders at week 30 within each group to a predefined minimum immunogenicity level of 50%; Test type: Other — The co-primary immunogenicity endpoint is analysed per arm, in a frequentist framework, in all randomised participants having received at least one vaccine administration and still HIV-negative at W30; p = 0.02, Binomial — One-sided test for the observed proportion being superior to the theoretical decision threshold of 50%

3. Secondary Outcome: To Assess the Tolerance of Each Prime-boost Combination
Description: Count of participants with at least one clinical/biological AE/SAE related to vaccine immunisation.
Time Frame: Between week 0 and week 52
Measure: Count of Participants; unit: Participants
Arm/Group | MVA HIV-B/LIPO-5 | LIPO-5/MVA HIV-B | GTU-MultiHIV B/LIPO-5 | GTU-MultiHIV B/MVA HIV-B
Number analyzed (Participants) | 23 | 23 | 23 | 23
Participants
  Clinical AE related to vaccine immunisation | 22 | 21 | 21 | 23
  Clinical SAE related to vaccine immunisation | 0 | 0 | 2 | 0
  Biological AE related to vaccine immunisation | 1 | 0 | 0 | 1
  Biological SAE related to vaccine immunisation | 1 | 0 | 0 | 1

4. Secondary Outcome: To Assess for Each Prime-boost Combination the Type of Vaccine-induced T Cell Response
Description: In all participants having received at least 1 dose of vaccine, the count of participants with HIV-specific ELISPOT response to at least one of stimulating HIV peptide pools.
Time Frame: At W2, W10 and W22 for reporting groups : MVA HIV-B/LIPO-5 and LIPO-5/MVA HIV-B. And at W2, W6, W14 and W22 for reporting groups : GTU-MultiHIV B/LIPO-T and GTU-MultiHIV B/MVA HIV-B.
Population: The number of participants differs due to the unavailability of some participants for some of the visits planned.
Measure: Count of Participants; unit: Participants
Groups:
- MVA HIV-B/LIPO-5: MVA HIV-B primes 0,5 mL IntraMmuscular at W0 and W8 LIPO-5 1mL IntraMuscular boosts at W20 and W28
Arm/Group | MVA HIV-B/LIPO-5 | LIPO-5/MVA HIV-B | GTU-MultiHIV B/LIPO-5 | GTU-MultiHIV B/MVA HIV-B
Number analyzed (Participants) | 23 | 23 | 23 | 23
Participants
  Week 2: number analyzed (Participants) | 22 | 20 | 22 | 22
  Week 2 | 5 | 1 | 1 | 1
  Week 6: number analyzed (Participants) | 0 | 0 | 21 | 19
  Week 6 |  |  | 0 | 1
  Week 10: number analyzed (Participants) | 22 | 22 | 0 | 0
  Week 10 | 13 | 1 |  |
  Week 14: number analyzed (Participants) | 0 | 0 | 20 | 21
  Week 14 |  |  | 0 | 0
  Week 22: number analyzed (Participants) | 20 | 20 | 20 | 20
  Week 22 | 9 | 8 | 1 | 12

ADVERSE EVENTS:
Time Frame: Each 92 participants were followed up for 52 weeks, unless they did not complete the study.
Arm/Group | MVA HIV-B/LIPO-5 | LIPO-5/MVA HIV-B | GTU-MultiHIV B/LIPO-5 | GTU-MultiHIV B/MVA HIV-B
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 3/23 | 5/23 | 7/23 | 3/23
Other Adverse Events (participants affected / at risk) | 22/23 | 23/23 | 22/23 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MVA HIV-B/LIPO-5 (N=23) | LIPO-5/MVA HIV-B (N=23) | GTU-MultiHIV B/LIPO-5 (N=23) | GTU-MultiHIV B/MVA HIV-B (N=23)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gilbert's syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitiligo (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine protein, quantitative (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Myelitis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eating disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MVA HIV-B/LIPO-5 (N=23) | LIPO-5/MVA HIV-B (N=23) | GTU-MultiHIV B/LIPO-5 (N=23) | GTU-MultiHIV B/MVA HIV-B (N=23)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LYMPHADENITIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 2 (2) | 1 (1)
MITRAL VALVE PROLAPSE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONJUNCTIVITIS (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OPHTHALMOPLEGIA (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ULCERATIVE KERATITIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (3) | 2 (2) | 3 (4) | 2 (2)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AGEUSIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANAL FISSURE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (3) | 1 (1)
DYSGEUSIA (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LIP DRY (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ASTHENIA (General disorders) | 6 (6) | 6 (11) | 9 (14) | 8 (12)
FACIAL PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 7 (9) | 4 (5) | 2 (6) | 9 (10)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 4 (5) | 1 (1) | 4 (4)
INJECTION SITE BRUISING (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
INJECTION SITE ERYTHEMA (General disorders) | 7 (10) | 5 (5) | 7 (10) | 6 (14)
INJECTION SITE GRANULOMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INJECTION SITE HAEMATOMA (General disorders) | 1 (1) | 2 (3) | 4 (4) | 3 (4)
INJECTION SITE HYPERSENSITIVITY (General disorders) | 7 (7) | 6 (10) | 6 (10) | 9 (11)
INJECTION SITE INDURATION (General disorders) | 5 (7) | 3 (3) | 7 (7) | 10 (15)
INJECTION SITE IRRITATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INJECTION SITE JOINT MOVEMENT IMPAIRMENT (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INJECTION SITE OEDEMA (General disorders) | 2 (2) | 1 (1) | 3 (3) | 2 (2)
INJECTION SITE PAIN (General disorders) | 21 (54) | 19 (39) | 17 (36) | 20 (56)
INJECTION SITE PARAESTHESIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INJECTION SITE PRURITUS (General disorders) | 2 (3) | 1 (1) | 2 (2) | 4 (5)
INJECTION SITE RASH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INJECTION SITE SWELLING (General disorders) | 3 (4) | 1 (1) | 0 (0) | 1 (1)
INJECTION SITE VESICLES (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NJECTION SITE OEDEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PUNCTURE SITE PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (3)
VESSEL PUNCTURE SITE HAEMATOMA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HAEMANGIOMA OF LIVER (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RHINITIS ALLERGIC (Immune system disorders) | 1 (1) | 3 (4) | 2 (2) | 0 (0)
RUBBER SENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
CONJUNCTIVITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CYSTITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EAR INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FOLLICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FURUNCLE (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GINGIVITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
HORDEOLUM (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
IMPETIGO (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFECTION PARASITIC (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MOLLUSCUM CONTAGIOSUM (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 2 (2) | 7 (8) | 6 (8) | 4 (4)
ORAL HERPES (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 2 (2)
PHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
RHINITIS (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 4 (4)
RHINOTRACHEITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (2)
SKIN BACTERIAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TINEA INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TINEA PEDIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
VAGINAL INFECTION (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
VIRAL PHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VIRAL RHINITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
BLOOD POTASSIUM DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLOOD URINE PRESENT (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
LIPASE INCREASED (Investigations) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
PROTEIN URINE PRESENT (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
TRANSAMINASES INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABNORMAL LOSS OF WEIGHT (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 3 (3) | 3 (5)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COCCYDYNIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LIGAMENT SPRAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
MUSCLE RIGIDITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 5 (9) | 3 (4) | 4 (5) | 11 (16)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TORTICOLLIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
FACIAL NEURALGIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GRAND MAL CONVULSION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 8 (9) | 7 (12) | 6 (8) | 11 (25)
HYPOAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
MIGRAINE WITH AURA (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
NERVE COMPRESSION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VERTIGO (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE STRESS DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
INSOMNIA (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
IRRITABILITY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SLEEP DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
STRESS (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
CALCULUS URINARY (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BREAST MASS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSMENORRHOEA (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 2 (3) | 1 (1)
EPIDIDYMITIS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
DERMATOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GENITAL RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PRURITUS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN DEPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CYST REMOVAL (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PILONIDAL SINUS REPAIR (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VARICOSE VEIN OPERATION (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VISION CORRECTION OPERATION (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HOT FLUSH (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PRESYNCOPE (Vascular disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
RAYNAUD'S PHENOMENON (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SYNCOPE (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results until their public communication.